CLINICAL TRIAL: NCT04595617
Title: Anti-αIIbβ3 Immunization in Glanzmann Thrombasthenia: Prevalence and Associated Risk Factors: Thrombasthenia Anti-αIIbβ3 Antibodies Study (TAAS)
Acronym: TAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/41
Record Dates: First submitted 2020-08-17; First posted 2020-10-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Glanzmann Thrombasthenia
Keywords: Glanzmann thrombasthenia; anti-GPIIb-IIIa immunization; MAIPA; Platelet transfusions; Recombinant activated factor VII
MeSH Terms: conditions — Thrombasthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diagnosis of Glanzmann Thrombastenia (GT) (Experimental): Antibodies screening will be systematically realized every six months (+/- 2 weeks) and after each last blood transfusion at 7-10 days and one month (+/- 2 weeks), during a period of 18 months
  Interventions: Biological: Antibodies screening

INTERVENTIONS:
Biological: Antibodies screening — All included GT patients will be enrolled from different national centres during a 6 months period. Antibodies screening will be systematically realized every six months (+/- 2 weeks) and after each last blood transfusion at 7-10 days and one month (+/- 2 weeks), during a period of 18 months.

SUMMARY:
This project aim to correlate risk factors (genetic, therapeutic and socio-demographic factors) to anti-αIIbβ3 antibodies formation following blood products transfusion (platelets or packed red cells) or pregnancy in a national cohort of GT patients.

DETAILED DESCRIPTION:
Glanzmann thrombasthenia (GT) is a rare autosomal recessive disorder caused by the absence or the dysfunction of the αIIbβ3 integrin, the most abundant receptor on platelets that mediates platelet aggregation through its binding of adhesive proteins. GT is readily identifiable by platelet function testing, and a lack of platelet aggregation in response to all physiological agonists is unique for this disease. The ITGA2B gene encodes for the αIIb subunit, whereas the ITGB3 gene encodes for β3. Mutations causing GT can affect either ITGA2B or ITGB3. The disease is characterized by spontaneous and trauma-related mucocutaneous bleeding, with variable expression ranging from easy bruising to fatal hemorrhages. Platelet transfusions are used to control or prevent life-threatening blood loss, but can become ineffective due to naturally occurring antibodies directed against αIIbβ3. Such antibodies are produced when patient's immune system comes into contact with normal αIIbβ3 expressing platelets.

There is no currently consensus concerning the frequency, the long-term evolution, or the formation of characteristics of antibodies from GT patients in relation to the nature of the defective gene (ITGA2B or ITGB3), gene variations or other factors. Research are needed to confirm that nature of the gene defect may have a causative role in antibody development. Moreover, strength and persistence of antibodies may vary among patients with the same mutation, suggesting that other factors, such as immune modifiers genes, play a role in shaping antibody repertoire.

Monoclonal antibody-specific immobilization of platelet antigens (MAIPA) is still considered as the reference method for evaluating the presence of anti-αIIbβ3 antibodies in GT patients. All the tests will be performed by the principal investigator site (Bordeaux).

ELIGIBILITY:
Inclusion Criteria:

* All patients with a clear diagnosis of Glanzmann Thrombastenia (GT), whatever the subtype of disease.
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant, or parents or legal representant for the child population, and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Current treatment that may interfere with anti-αIIbβ3 antibodies detection, such as intravenous immunoglobulins within the previous month.
* Psychiatric, social or behavioral condition judged to be non-compatible with the respect of the protocol, including good observance of treatment and compliance to follow-up.
* Adult protected by the law.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Characterization of change of an anti-αIIbβ3 immunization | From inclusion to 18 months visit
  Characterization of change of an anti-αIIbβ3 immunization will be assessed with Indirect MoAb-specific immobilization of platelet antigens (MAIPA)
Number of patients with positive anti-αIIbβ3 antibodies in relation to risk factors | From inclusion to 18 months visit
  Risk factors could be subtype of GT, year of birth, ITGA2B or ITGB3 gene mutation

SECONDARY OUTCOMES:
Determination of the prevalence of anti-αIIbβ3 antibodies in a regional cohort of GT patients | From inclusion to 18 months visit
  Presence of anti-αIIbβ3 antibodies will be assessed with Indirect MoAb-specific immobilization of platelet antigens (MAIPA)
Description of the kinetic of an anti-αIIbβ3 immunization following blood transfusion | At 7-10 days and 1 month (+/-2 weeks) after each blood transfusion
  Repetition of the antibodies measurements with Indirect MoAb-specific immobilization of platelet antigens (MAIPA)
Determination of the mechanism of anti-αIIbβ3 antibodies blocking integrin function by determining the capacity of anti-αIIbβ3 antibodies to impair fibrinogen binding | through study completion, an average of 2 years
  In vitro studies will be performed by mixing serum of patients with washed donors' platelets and inhibition of the integrin will be studied by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu FIORE, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CHU Bordeaux - Hôpital Haut-Lévêque, Bordeaux
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital Bicêtre, APHP, Le Kremlin-Bicêtre
  - Hôpital la Timone, APHM, Marseille
  - CHU Nîmes, Nîmes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No